CLINICAL TRIAL: NCT03534011
Title: Resuscitative Balloon Occlusion of the Aorta (REBOA) in Non-traumatic Out of Hospital Cardiac Arrest - a Pilot Study
Brief Title: Resuscitative Balloon Occlusion of the Aorta in Non-traumatic Out of Hospital Cardiac Arrest
Acronym: REBOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Norwegian Air Ambulance Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/51
Record Dates: First submitted 2018-05-12; First posted 2018-05-23 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Balloon occlusion; Air ambulances; Aorta; Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REBOA (Experimental): Resuscitative Balloon Occlusion of the Aorta after advanced cardiac life support if return of spontaneous circulation is not achieved
  Interventions: Procedure: Resuscitative Balloon Occlusion of the Aorta; Device: REBOA catheter

INTERVENTIONS:
Procedure: Resuscitative Balloon Occlusion of the Aorta — If return of spontaneous circulation (ROSC) is not achieved after advanced cardiac life support (ACLS) is established, a REBOA catheter is inserted via the femoral artery and the aortic balloon inflated, according to a procedure described in a separate document. Ultrasound is used to limit risk related to cannulation and placement of the guidewire.
  Other Names: REBOA
Device: REBOA catheter — Catheter with a Resuscitative Balloon for Occlusion of the Aorta

SUMMARY:
The primary aim of this study is to investigate the feasibility and complications of inserting a REBOA-catheter to patients suffering from non-traumatic out-of-hospital cardiac arrest, by anesthesiologist working in the pre-hospital setting. The study will include patients in the catchment population of St. Olavs University Hospital, Trondheim area, Norway. The REBOA technique (resuscitative balloon occlusion of the aorta) is a well-known treatment used on other indications, both in-hospital and pre-hospital. It has also been utilized in several animal studies on non-traumatic cardiac arrest and has shown to augment myocardial and cerebral perfusion during cardio-pulmonary resuscitation. There are no systematic studies on humans with REBOA in non-traumatic cardiac arrest. The study will also investigate the time needed to perform a REBOA procedure in cardiac arrest patients receiving advanced cardiac life support. This additional treatment might contribute to increase the survival rate of cardiac arrest patients.

DETAILED DESCRIPTION:
If return of spontaneous circulation (ROSC) is not achieved after advanced cardiac life support (ACLS as described in the present guidelines from the Norwegian Resuscitation Council) is established, a REBOA catheter is inserted via the femoral artery and the aortic balloon inflated, according to a procedure described in a separate document. Ultrasound is used to limit risk related to cannulation and placement of the guidewire. The ultrasound images will be stored and later processed by the principal investigator. If the physician experiences technical problems during the procedure (i.e. severe difficulties in establishing vascular access, resistance during insertion of the guidewire, introducer or balloon catheter, severe bleeding, prolonged time consumption) the effort will be aborted. If ROSC is achieved, the aortic balloon is deflated gently. If the patient re-enters cardiac arrest, the normal ACLS-guideline is followed. The balloon is then re-inflated, as described in the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Non-traumatic cardiac arrest
* Witnessed cardiac arrest
* Less than 10 minutes from observed cardiac arrest to start of basic or advanced cardiac life support (BCLS/ACLS)

Exclusion Criteria:

* Traumatic cardiac arrest, including patients rescued from avalanches
* Hypothermic patients, including drowning
* Pregnancy
* End-stage terminal illness
* Suspected neurologic injury as the etiology of the arrest
* Strangulations
* Other factors as decided by the treating physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility | 20 minutes
  Report of the feasibility is based on the ease of performing the REBOA procedure. A checklist which grades the different technical moments and time consumption of the procedure is described in a separate document. All physicians will be interviewed by the principal investigator to assess other factors that influenced the in-field performance of the procedure (i.e weather, temperature, light condition, body habitus, constrained room)
Complications | 30 days
  Complications related to the REBOA procedure, immediate or late, as well as negative interaction on the cardiopulmonary resuscitation (CPR)

CONTACTS AND LOCATIONS:
Overall Officials: Sindre Mellesmo, md, Study Director — St. Olavs Hospital; Jostein Rødseth Brede, md, Principal Investigator — St. Olavs Hospital
Locations (1):
- Trondheim area, Trondheim, Norway

REFERENCES:
- [Background] Brede JR, Lafrenz T, Kruger AJ, Sovik E, Steffensen T, Kriesi C, Steinert M, Klepstad P. Resuscitative endovascular balloon occlusion of the aorta (REBOA) in non-traumatic out-of-hospital cardiac arrest: evaluation of an educational programme. BMJ Open. 2019 May 9;9(5):e027980. doi: 10.1136/bmjopen-2018-027980. PMID 31076474
- [Background] Brede JR, Lafrenz T, Klepstad P, Skjaerseth EA, Nordseth T, Sovik E, Kruger AJ. Feasibility of Pre-Hospital Resuscitative Endovascular Balloon Occlusion of the Aorta in Non-Traumatic Out-of-Hospital Cardiac Arrest. J Am Heart Assoc. 2019 Nov 19;8(22):e014394. doi: 10.1161/JAHA.119.014394. Epub 2019 Nov 11. PMID 31707942
- [Result] Brede JR, Skjaerseth E, Klepstad P, Nordseth T, Kruger AJ. Changes in peripheral arterial blood pressure after resuscitative endovascular balloon occlusion of the aorta (REBOA) in non-traumatic cardiac arrest patients. BMC Emerg Med. 2021 Dec 15;21(1):157. doi: 10.1186/s12873-021-00551-y. PMID 34911463